CLINICAL TRIAL: NCT04201093
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, 27-Week Trial to Evaluate the Efficacy, Safety, and Tolerability of Two Fixed Doses of Tavapadon in Early Parkinson's Disease (TEMPO-1 TRIAL)
Brief Title: Fixed-Dose Trial in Early Parkinson's Disease (PD)
Acronym: TEMPO-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVL-751-PD-001; 2019-002949-38 (EudraCT Number)
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: Parkinsonian Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Tavapadon 5 mg (Experimental): Participants will receive tavapadon tablet titrated up to 5 milligram (mg) once daily (QD) orally for 27 weeks.
  Interventions: Drug: Tavapadon
- Tavapadon 15 mg (Experimental): Participants will receive tavapadon tablet titrated up to 15 milligram (mg) QD orally for 27 weeks.
  Interventions: Drug: Tavapadon
- Placebo (Placebo Comparator): Participants will receive placebo matching to tavapadon tablet QD orally for 27 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tavapadon — Participants will be randomized to receive tavapadon 5mg tablet once daily orally for 27 weeks.
  Other Names: PF-06649751; CVL-751
  Arms: Tavapadon 5 mg
Drug: Placebo — Participants will receive placebo matching to tavapadon QD orally for 27 weeks.
  Arms: Placebo
Drug: Tavapadon — Participants will be randomized to receive tavapadon 15mg tablet once daily orally for 27 weeks.
  Other Names: PF-06649751; CVL-751
  Arms: Tavapadon 15 mg

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy, safety and pharmacokinetics (PK) of 2 fixed doses of tavapadon and placebo in participants with early PD.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female participants aged 40 to 80 years, inclusive, at the time of signing the informed consent form (ICF)
* Sexually active men or women of childbearing potential must agree to use acceptable (at minimum) or highly effective birth control, or remain abstinent during the trial and for 4 weeks after the last dose of trial treatment
* Participants who are capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in the protocol
* Participants with a diagnosis of PD that is consistent with the UK Parkinson's Disease Society Brain Bank diagnostic criteria
* Participants with modified Hoehn and Yahr stage 1, 1.5, or 2
* Participants with disease duration (from time of diagnosis) of less than (<) 3 years and disease progression in the 3 years before signing the ICF
* Participants with an MDS-UPDRS Part II score >=2 and Part III score >=10 at the Screening Visit and at the Baseline Visit
* Participants with early PD who, in the opinion of the investigator, require pharmacologic intervention for disease management
* Participants who are treatment naïve or have a history of prior incidental treatment with dopaminergic agents (including Levodopa [L-Dopa] and dopamine receptor agonist medications) for <3 months in total but not within 2 months of the Baseline Visit. Prior and concurrent use of monoamine oxidase B (MAO-B) inhibitors is permitted if use was initiated >90 days before the Baseline Visit and the dosage will remain stable for the duration of the trial (i.e, no change in the MAO-B inhibitor dose is permitted during the trial)
* Participants who are willing and able to refrain from any PD medications that are not permitted by the protocol (including dopaminergic agents) throughout participation in the trial.

Key Exclusion Criteria:

* Participants with a history or clinical features consistent with essential tremor, atypical or secondary parkinsonian syndrome (including, but not limited to, progressive supra nuclear palsy, multiple system atrophy, cortico-basal degeneration, or drug-induced or post stroke parkinsonism).
* Participants with a history of nonresponse or insufficient response to L-Dopa at therapeutic dosages.
* Participants with a history or current diagnosis of a clinically significant impulse control disorder (Disruptive, Impulse Control, and Conduct Disorder per DSM-5).
* Participants with the presence of or history of brain tumor, hospitalization for severe head trauma, epilepsy (as defined by the International League Against Epilepsy), or seizures.
* Participants with a history of psychosis or hallucinations within the previous 12 months.
* Participants who answer "yes" on the Columbia-Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation Item 4 or Item 5 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan, or Active Suicidal Ideation with Specific Plan and Intent) and whose most recent episode meeting the criteria for C-SSRS Item 4 or Item 5 occurred within the last 6 months, OR Participants who answer "yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) and whose most recent episode meeting the criteria for any of these 5 C-SSRS Suicidal Behavior Items occurred within the last 2 years, OR Participants who, in the opinion of the investigator, present a serious risk of suicide.
* Participants with substance abuse or dependence disorder, including alcohol, benzodiazepines, and opioids, but excluding nicotine, within the past 6 months (180 days)
* Participants with dementia or cognitive impairment that, in the judgement of the investigator, would exclude the participant from understanding the ICF or participating in the trial
* Participants with any condition that could possibly affect drug absorption, including bowel resections, bariatric weight loss surgery, or gastrectomy (this does not include gastric banding).
* Participants who have a positive result for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV) antibodies at screening.
* Participants with a history of myocardial infarction with residual atrial, nodal, or ventricular arrhythmias that are not controlled with medical and/or surgical intervention; second- or third-degree atrioventricular block; sick sinus syndrome; severe or unstable angina; or congestive heart failure within the last 12 months. A recent (less than or equal to [<=] 12 months) history of myocardial infarction with secondary arrhythmias is exclusionary regardless of the therapeutic control.
* Participants with a history of neuroleptic malignant syndrome.
* Participants who are currently receiving moderate or strong CYP3A4 inducers or CYP3A4 inhibitors (except for topical administration).
* Participants with a positive urine drug screen for illicit drugs are excluded and may not be retested or rescreened. Participants with a positive urine drug screen resulting from use of marijuana (any Tetrahydrocannabinol [THC]-containing product), prescription, or over-the-counter medications or products that, in the investigator's documented opinion, do not signal a clinical condition that would impact the safety of the participant or interpretation of the trial results may continue evaluation for the trial following consultation and approval by the medical monitor
* Participants with a Montreal Cognitive Assessment (MoCA) score <26
* Participants with clinically significant orthostatic hypotension (eg, syncope)
* Participants with a 12-lead ECG demonstrating a QTcF interval >450 msec
* Participants with moderate or severe renal impairment (creatinine clearance as estimated by Cockcroft-Gault formula <30 mL/min or on dialysis)
* Participants with any of the following abnormalities in clinical laboratory tests at the Screening Visit, as assessed by the central laboratory and confirmed by a single repeat measurement, if deemed necessary:

  * Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) >=3 × Upper Limit Normal (ULN).
  * Total bilirubin >=1.5 × ULN. Participants with a history of Gilbert's syndrome may be eligible provided they have a value <ULN for direct bilirubin.
* Participants with other abnormal laboratory test results, vital sign results, or ECG findings unless, in the judgment of the investigator, the findings are not medically significant and would not impact the safety of the participants or the interpretation of the trial results.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., MD, Study Director — AbbVie
Locations (72):
- United States (27):
  - Birmingham, Alabama, Birmingham, Alabama
  - Little Rock, Arkansas, Little Rock, Arkansas
  - Fountain Valley, California, Fountain Valley, California
  - Los Angeles, California, Los Angeles, California
  - Pasadena, California, Pasadena, California
  - Englewood, Colorado, Englewood, Colorado
  - Adventura, Florida, Adventura, Florida
  - Boca Raton, Florida, Boca Raton, Florida
  - Tampa, Florida, Tampa, Florida
  - Augusta, Georgia, Augusta, Georgia
  - Savannah, Georgia, Savannah, Georgia
  - Chicago, Illinois, Chicago, Illinois
  - Kansas City, Kansas, Kansas City, Kansas
  - Scarborough, Maine, Scarborough, Maine
  - Boston, Massachusetts, Boston, Massachusetts
  - East Lansing, Michigan, East Lansing, Michigan
  - Las Vegas, Nevada, Las Vegas, Nevada
  - Asheville, North Carolina, Asheville, North Carolina
  - Durham, North Carolina, Durham, North Carolina
  - Columbus, Ohio, Columbus, Ohio
  - Toledo, Ohio, Toledo, Ohio
  - Philadelphia, Pennsylvania, Philadelphia, Pennsylvania
  - Georgetown, Texas, Georgetown, Texas
  - Houston, Texas, Houston, Texas
  - Lubbock, Texas, Lubbock, Texas
  - Burlington, Vermont, Burlington, Vermont
  - Virginia Beach, Virginia, Virginia Beach, Virginia
- Australia (3):
  - Erina, New South Wales, Erina, New South Wales
  - Woolloongabba, Queensland, Woolloongabba, Queensland
  - Parkville, Victoria, Parkville, Victoria
- Bulgaria (6):
  - Medical center VITA1, Pleven, Pleven
  - Pleven, Bulgaria, Pleven
  - Pleven, Pleven
  - Multiprofile Hospital, Sofia, Sofia
  - Sofia, Sofia
  - DCC Neoclinic, Sofia
- Canada (2):
  - Ottawa, Ontario, Ottawa, Ontario
  - Toronto, Ontario, Toronto, Ontario
- Czechia (3):
  - Poliklinika, Chocen,, Choceň, Chocen
  - Prague,, Prague
  - Rychnov nad Kněžnou, Rychnov nad Kněžnou
- France (5):
  - Creteil, Créteil, Creteil
  - Boulevard Pinel, Bron, Bron
  - Grenoble cedex, Grenoble
  - Nancy, France, Nancy
  - Nîmes cedex, Nîmes
- Germany (5):
  - Muenster, Münster, Muenster
  - Bad Homburg, Bad Homburg
  - Duesseldorf,, Düsseldorf
  - Haag in Oberbayern, Haag in Oberbayern
  - Stadtroda, Stadtroda
- Israel (4):
  - Haifa, Haifa
  - Petah Tiqva, Petah Tikva
  - Ramat Gan, Ramat Gan
  - Tel Aviv, Tel Aviv
- Italy (4):
  - Milano, Milan
  - Padova, Padua
  - Pisa, Pisa
  - Rome, Rome
- Poland (3):
  - Kraków, Krakow
  - Singua, Warsaw
  - Lodz, Lodz, Łódź Voivodeship
- Spain (6):
  - Elche, Elche, Alicante
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Madrid, Spain, Madrid
  - Terrassa, Terrassa
  - Valencia, Valencia
- Ukraine (4):
  - Zaporiizhzhya, Zaporizhzhya, Zaporiizhzhya
  - Zaporozhya, Zaporizhzhya, Zaporozhya
  - Dnipro, Dnipro
  - Kharkiv, Kharkiv

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this Phase 3, Double-Blind study, a total of 529 subjects with Parkinson's Disease (PD) were randomized in a 1:1:1 ratio to 3 treatment groups: Tavapadon 5 mg, Tavapadon 15 mg, or Placebo once daily (QD) for 27 Weeks.
Groups:
- Placebo: Participants will receive placebo matching to tavapadon tablet once daily once daily (QD) orally for 27 weeks.
- Tavapadon 5 mg: Participants will receive tavapadon tablet titrated up to 5 milligram (mg) QD orally for 27 weeks.
Period: Overall Study
Arm/Group | Placebo | Tavapadon 5 mg | Tavapadon 15 mg
Started | 175 | 177 | 177
Completed | 148 | 134 | 118
Not Completed | 27 | 43 | 59
Not completed — Adverse Event | 6 | 29 | 35
Not completed — Death | 2 | 1 | 0
Not completed — Lack of Efficacy | 5 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Failure to Meet Continuation Criteria | 0 | 0 | 1
Not completed — Treatment with Prohibited Concomitant Medications | 0 | 0 | 1
Not completed — Non-Compliance with Study Schedule | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0
Not completed — Site Terminated by Sponsor | 5 | 3 | 1
Not completed — Withdrawal by Subject | 7 | 8 | 15
Not completed — Other | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Includes all enrolled subjects that received at least one dose of study drug.
Groups:
- Placebo: Participants will receive placebo matching to tavapadon tablet once daily (QD) orally for 27 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Tavapadon 5 mg | Tavapadon 15 mg | Total
Number analyzed (Participants) | 175 | 177 | 177 | 529
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (9.62) | 63.7 (9.80) | 63.8 (9.40) | 63.7 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 66 | 58 | 187
  Male | 112 | 111 | 119 | 342
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 13 | 10 | 32
  Not Hispanic or Latino | 154 | 153 | 158 | 465
  Unknown or Not Reported | 12 | 11 | 9 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 3 | 0 | 2 | 5
  White | 168 | 174 | 172 | 514
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 2 | 5
MDS-UPDRS Score at Baseline (Parts II and III Combined) [Mean (Standard Deviation); unit: units on a scale] — The MDS-UPDRS rating tool was used to follow longitudinal course of Parkinson's Disease and consisted of 4 parts.Part 1:Non-motor aspects of experiences of daily living[13 items,Score range(SR):0-52];Part 2:Motor aspects of experiences of daily living(13 items,SR:0-52);Part 3:Motor examination(18 items,SR:0-132);Part 4:Motor complications(6 items,SR:0-24.Not collected).Each item has 0-4 rating on scale from 0(normal)-4(severe).Higher values represent a worse outcome.Parts 2 and 3 combined is the sum of Part 2 and Part 3 scores at each assessment time for each participant(31 items,SR:0-184).
  units on a scale | 32.0 (9.96) | 31.3 (10.87) | 32.1 (11.55) | 31.8 (10.80)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the MDS-UPDRS Parts II and III Combined Score
Description: The Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) rating tool was used to follow longitudinal course of Parkinson's Disease. It was made up of 4 parts: Part 1: Non-motor aspects of experiences of daily living (13 items. Score range: 0-52); Part 2: Motor aspects of experiences of daily living (13 items. Score range: 0-52); Part 3: Motor examination (18 items. Score range: 0-132); Part 4: Motor complications (6 items. Score range: 0-24. Part 4 was not collected in this trial). Each item has 0-4 rating on scale from 0 (normal) to 4 (severe). Higher values represent a worse outcome. A negative change from baseline represents an improvement in motor function. Parts 2 and 3 combined is the sum of Part 2 score and Part 3 score at each assessment time for each participant. The combined score assesses 31 items with score range: 0-184.
Time Frame: Week 26
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Tavapadon 5 mg | Tavapadon 15 mg
Number analyzed (Participants) | 148 | 132 | 116
score on a scale | 1.8 (0.82) | -9.7 (0.86) | -10.2 (0.88)
Statistical Analysis 1: Comparison: Placebo vs Tavapadon 5 mg; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — LS Means, SE, difference from placebo, and CI's are estimated using a mixed effects repeated measures model with fixed effects for treatment group, visits, treatment by visit interaction and MAO-B inhibitor use with the baseline value as a covariate; LS Mean of Difference = -11.5, 95% CI 2-sided [-13.8 to -9.2], Standard Error of Mean 1.16
Statistical Analysis 2: Comparison: Placebo vs Tavapadon 15 mg; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -12.1, 95% CI 2-sided [-14.4 to -9.8], Standard Error of Mean 1.17

2. Secondary Outcome: Change From Baseline in the MDS-UPDRS Part II Score
Description: The Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) rating tool was used to follow longitudinal course of Parkinson's Disease. It was made up of 4 parts: Part 1: Non-motor aspects of experiences of daily living (13 items. Score range: 0-52); Part 2: Motor aspects of experiences of daily living (13 items. Score range: 0-52); Part 3: Motor examination (18 items. Score range: 0-132); Part 4: Motor complications (6 items. Score range: 0-24. Part 4 was not collected in this trial). Each item has 0-4 rating on scale from 0 (normal) to 4 (severe). Higher values represent a worse outcome. A negative change from baseline represents an improvement in motor function.
Time Frame: Week 26
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Tavapadon 5 mg | Tavapadon 15 mg
Number analyzed (Participants) | 148 | 132 | 116
score on a scale | 0.9 (0.30) | -1.6 (0.31) | -1.7 (0.32)
Statistical Analysis 1: Comparison: Placebo vs Tavapadon 5 mg; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -2.5, 95% CI 2-sided [-3.3 to -1.7], Standard Error of Mean 0.43
Statistical Analysis 2: Comparison: Placebo vs Tavapadon 15 mg; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -2.6, 95% CI 2-sided [-3.4 to -1.7], Standard Error of Mean 0.43

3. Secondary Outcome: Percentage of Responders With a Score of "Much Improved" or "Very Much Improved" on PGIC
Description: The Patient Global Impression of Change (PGIC) is a 7-point response scale. The participant response to the question, "Compared to your condition at the beginning of treatment, how much has your condition changed?" was assessed. Scores ranged from 1-7 on a scale of 1 (very much improved) to 7 (very much worse). Higher values represent a worse outcome.
Time Frame: Week 26
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tavapadon 5 mg | Tavapadon 15 mg
Number analyzed (Participants) | 147 | 132 | 117
Participants | 18 | 60 | 52
Statistical Analysis 1: Comparison: Placebo vs Tavapadon 5 mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Odds Ratio (OR) = 6.148, 95% CI 2-sided [3.339 to 11.321]
Statistical Analysis 2: Comparison: Placebo vs Tavapadon 15 mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Odds Ratio (OR) = 5.968, 95% CI 2-sided [3.220 to 11.062]

4. Secondary Outcome: Change From Baseline in the MDS-UPDRS Parts II and III Combined Score
Description: as for outcome 1
Time Frame: Week 5, 8, 11, 14, 18, 22, 26, and 27
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Tavapadon 5 mg | Tavapadon 15 mg
Number analyzed (Participants) | 174 | 174 | 172
score on a scale
  Week 5: number analyzed (Participants) | 171 | 154 | 159
  Week 5 | -1.2 (0.57) | -4.4 (0.59) | -4.7 (0.59)
  Week 8: number analyzed (Participants) | 168 | 147 | 150
  Week 8 | -2.2 (0.62) | -6.9 (0.65) | -6.7 (0.65)
  Week 11: number analyzed (Participants) | 160 | 138 | 135
  Week 11 | -0.9 (0.72) | -8.1 (0.75) | -9.1 (0.75)
  Week 14: number analyzed (Participants) | 158 | 142 | 134
  Week 14 | -1.2 (0.74) | -8.8 (0.78) | -9.4 (0.78)
  Week 18: number analyzed (Participants) | 153 | 138 | 129
  Week 18 | 0.4 (0.78) | -9.1 (0.82) | -9.7 (0.83)
  Week 22: number analyzed (Participants) | 150 | 137 | 126
  Week 22 | 0.4 (0.81) | -9.6 (0.84) | -10.9 (0.86)
  Week 26: number analyzed (Participants) | 148 | 132 | 116
  Week 26 | 1.8 (0.82) | -9.7 (0.86) | -10.2 (0.88)
  Week 27: number analyzed (Participants) | 148 | 134 | 119
  Week 27 | 2.2 (0.92) | -8.6 (0.96) | -10.0 (0.99)
Statistical Analysis 1: Comparison: Placebo vs Tavapadon 5 mg; Week 26; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -11.5, 95% CI 2-sided [-13.8 to -9.2], Standard Error of Mean 1.16
Statistical Analysis 2: Comparison: Placebo vs Tavapadon 15 mg; Week 26; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -12.1, 95% CI 2-sided [-14.4 to -9.8], Standard Error of Mean 1.17

5. Secondary Outcome: Change From Baseline in the MDS-UPDRS Parts I, II and III Combined Score
Description: The Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) rating tool was used to follow longitudinal course of Parkinson's Disease. It was made up of 4 parts: Part 1: Non-motor aspects of experiences of daily living (13 items. Score range: 0-52); Part 2: Motor aspects of experiences of daily living (13 items. Score range: 0-52); Part 3: Motor examination (18 items. Score range: 0-132); Part 4: Motor complications (6 items. Score range: 0-24. Part 4 was not collected in this trial). Each item has 0-4 rating on scale from 0 (normal) to 4 (severe). Higher values represent a worse outcome. A negative change from baseline represents an improvement in motor function. Parts 1, 2, and 3 combined is the sum of Part 1, Part 2, and Part 3 scores at each assessment time for each participant. The combined score assesses 44 items with score range: 0-236.
Time Frame: Week 5, 8, 11, 14, 18, 22, 26, and 27
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Tavapadon 5 mg | Tavapadon 15 mg
Number analyzed (Participants) | 174 | 174 | 172
score on a scale
  Week 5: number analyzed (Participants) | 171 | 154 | 159
  Week 5 | -1.2 (0.67) | -3.9 (0.69) | -4.0 (0.69)
  Week 8: number analyzed (Participants) | 168 | 147 | 150
  Week 8 | -2.6 (0.72) | -6.4 (0.76) | -6.2 (0.75)
  Week 11: number analyzed (Participants) | 160 | 138 | 135
  Week 11 | -1.2 (0.81) | -7.7 (0.86) | -8.6 (0.86)
  Week 14: number analyzed (Participants) | 158 | 142 | 134
  Week 14 | -1.5 (0.85) | -8.8 (0.89) | -8.7 (0.90)
  Week 18: number analyzed (Participants) | 153 | 138 | 129
  Week 18 | 0.3 (0.91) | -9.3 (0.95) | -9.1 (0.96)
  Week 22: number analyzed (Participants) | 150 | 137 | 126
  Week 22 | 0.2 (0.94) | -9.5 (0.98) | -10.3 (1.00)
  Week 26: number analyzed (Participants) | 148 | 132 | 116
  Week 26 | 2.3 (0.95) | -9.4 (1.00) | -9.7 (1.02)
  Week 27: number analyzed (Participants) | 148 | 134 | 119
  Week 27 | 2.4 (1.06) | -8.5 (1.11) | -9.4 (1.14)
Statistical Analysis 1: Comparison: Placebo vs Tavapadon 5 mg; Week 26; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -11.7, 95% CI 2-sided [-14.4 to -9.1], Standard Error of Mean 1.35
Statistical Analysis 2: Comparison: Placebo vs Tavapadon 15 mg; Week 26; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -12.0, 95% CI 2-sided [-14.7 to -9.3], Standard Error of Mean 1.37

6. Secondary Outcome: Change From Baseline in the MDS-UPDRS Parts I, II and III Individual Score
Description: as for outcome 2
Time Frame: Week 5, 8, 11, 14, 18, 22, 26, and 27
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Tavapadon 5 mg | Tavapadon 15 mg
Number analyzed (Participants) | 174 | 174 | 172
score on a scale
  Part I: Week 5: number analyzed (Participants) | 171 | 155 | 160
  Part I: Week 5 | 0.0 (0.23) | 0.6 (0.24) | 0.7 (0.24)
  Part I: Week 8: number analyzed (Participants) | 168 | 149 | 151
  Part I: Week 8 | -0.4 (0.23) | 0.5 (0.24) | 0.4 (0.24)
  Part I: Week 11: number analyzed (Participants) | 161 | 141 | 135
  Part I: Week 11 | -0.3 (0.23) | 0.4 (0.24) | 0.4 (0.25)
  Part I: Week 14: number analyzed (Participants) | 158 | 142 | 134
  Part I: Week 14 | -0.2 (0.25) | 0.0 (0.27) | 0.6 (0.27)
  Part I: Week 18: number analyzed (Participants) | 153 | 138 | 129
  Part I: Week 18 | -0.1 (0.25) | -0.2 (0.26) | 0.5 (0.27)
  Part I: Week 22: number analyzed (Participants) | 150 | 137 | 126
  Part I: Week 22 | -0.2 (0.26) | 0.2 (0.27) | 0.4 (0.28)
  Part I: Week 26: number analyzed (Participants) | 148 | 132 | 116
  Part I: Week 26 | 0.5 (0.27) | 0.2 (0.28) | 0.4 (0.29)
  Part I: Week 27: number analyzed (Participants) | 148 | 134 | 119
  Part I: Week 27 | 0.2 (0.27) | 0.2 (0.28) | 0.3 (0.29)
  Part II: Week 5: number analyzed (Participants) | 171 | 155 | 160
  Part II: Week 5 | -0.2 (0.22) | -0.8 (0.23) | -1.0 (0.22)
  Part II: Week 8: number analyzed (Participants) | 168 | 149 | 151
  Part II: Week 8 | -0.5 (0.23) | -1.0 (0.25) | -1.6 (0.24)
  Part II: Week 11: number analyzed (Participants) | 161 | 141 | 135
  Part II: Week 11 | 0.0 (0.26) | -1.7 (0.27) | -2.0 (0.27)
  Part II: Week 14: number analyzed (Participants) | 159 | 142 | 134
  Part II: Week 14 | -0.1 (0.27) | -1.6 (0.28) | -2.0 (0.28)
  Part II: Week 18: number analyzed (Participants) | 153 | 138 | 129
  Part II: Week 18 | 0.4 (0.29) | -1.9 (0.31) | -1.8 (0.31)
  Part II: Week 22: number analyzed (Participants) | 150 | 137 | 126
  Part II: Week 22 | 0.3 (0.28) | -1.7 (0.29) | -2.1 (0.29)
  Part II: Week 26: number analyzed (Participants) | 148 | 132 | 116
  Part II: Week 26 | 0.9 (0.30) | -1.6 (0.31) | -1.7 (0.32)
  Part II: Week 27: number analyzed (Participants) | 148 | 134 | 119
  Part II: Week 27 | 0.9 (0.31) | -1.7 (0.32) | -1.8 (0.33)
  Part III: Week 5: number analyzed (Participants) | 171 | 154 | 160
  Part III: Week 5 | -1.0 (0.44) | -3.7 (0.46) | -3.7 (0.45)
  Part III: Week 8: number analyzed (Participants) | 168 | 147 | 150
  Part III: Week 8 | -1.7 (0.50) | -6.0 (0.52) | -5.1 (0.52)
  Part III: Week 11: number analyzed (Participants) | 160 | 138 | 135
  Part III: Week 11 | -1.0 (0.55) | -6.5 (0.58) | -7.1 (0.59)
  Part III: Week 14: number analyzed (Participants) | 158 | 142 | 134
  Part III: Week 14 | -1.1 (0.58) | -7.2 (0.61) | -7.4 (0.61)
  Part III: Week 18: number analyzed (Participants) | 153 | 138 | 129
  Part III: Week 18 | 0.0 (0.60) | -7.3 (0.63) | -7.9 (0.64)
  Part III: Week 22: number analyzed (Participants) | 150 | 137 | 126
  Part III: Week 22 | 0.0 (0.64) | -8.0 (0.67) | -8.8 (0.68)
  Part III: Week 26: number analyzed (Participants) | 148 | 132 | 116
  Part III: Week 26 | 0.9 (0.63) | -8.1 (0.66) | -8.5 (0.68)
  Part III: Week 27: number analyzed (Participants) | 148 | 134 | 119
  Part III: Week 27 | 1.1 (0.71) | -7.1 (0.75) | -8.3 (0.77)
Statistical Analysis 1: Comparison: Placebo vs Tavapadon 5 mg; Part I: Week 26; Test type: Superiority; p = 0.4822, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.3, 95% CI 2-sided [-1.0 to 0.5], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: Placebo vs Tavapadon 15 mg; Part I: Week 26; Test type: Superiority; p = 0.7742, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.1, 95% CI 2-sided [-0.9 to 0.6], Standard Error of Mean 0.38
Statistical Analysis 3: Comparison: Placebo vs Tavapadon 5 mg; Part II: Week 26; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -2.5, 95% CI 2-sided [-3.3 to -1.7], Standard Error of Mean 0.43
Statistical Analysis 4: Comparison: Placebo vs Tavapadon 15 mg; Part II: Week 26; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -2.6, 95% CI 2-sided [-3.4 to -1.7], Standard Error of Mean 0.43
Statistical Analysis 5: Comparison: Placebo vs Tavapadon 5 mg; Part III: Week 26; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -9.0, 95% CI 2-sided [-10.8 to -7.3], Standard Error of Mean 0.89
Statistical Analysis 6: Comparison: Placebo vs Tavapadon 15 mg; Part III: Week 26; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -9.4, 95% CI 2-sided [-11.2 to -7.6], Standard Error of Mean 0.90

7. Secondary Outcome: Change From Baseline in the CGI-S Score
Description: The Global Impression - Severity of Illness (CGI-S) Score is a clinician's impression of a participant's severity of illness on a 7-point scale. Scores ranged from 1-7 on a scale of 1 (normal) to 7 (among the most extremely ill participants). Higher values represent a worse outcome.
Time Frame: Week 5, 8, 11, 14, 18, 22, 26, and 27
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Tavapadon 5 mg | Tavapadon 15 mg
Number analyzed (Participants) | 174 | 174 | 172
score on a scale
  Week 5: number analyzed (Participants) | 171 | 155 | 160
  Week 5 | 0.0 (0.04) | -0.1 (0.05) | 0.0 (0.05)
  Week 8: number analyzed (Participants) | 168 | 148 | 151
  Week 8 | 0.0 (0.05) | -0.1 (0.05) | -0.1 (0.05)
  Week 11: number analyzed (Participants) | 161 | 141 | 135
  Week 11 | 0.0 (0.05) | -0.2 (0.05) | -0.3 (0.05)
  Week 14: number analyzed (Participants) | 158 | 141 | 133
  Week 14 | 0.1 (0.05) | -0.2 (0.05) | -0.3 (0.05)
  Week 18: number analyzed (Participants) | 153 | 138 | 129
  Week 18 | 0.1 (0.05) | -0.3 (0.06) | -0.3 (0.06)
  Week 22: number analyzed (Participants) | 150 | 137 | 126
  Week 22 | 0.1 (0.05) | -0.2 (0.06) | -0.3 (0.06)
  Week 26: number analyzed (Participants) | 148 | 132 | 117
  Week 26 | 0.2 (0.05) | -0.3 (0.05) | -0.2 (0.06)
  Week 27: number analyzed (Participants) | 147 | 134 | 119
  Week 27 | 0.1 (0.05) | -0.2 (0.06) | -0.2 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Tavapadon 5 mg; Week 26; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.5, 95% CI 2-sided [-0.6 to -0.3], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Placebo vs Tavapadon 15 mg; Week 26; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.4, 95% CI 2-sided [-0.5 to -0.2], Standard Error of Mean 0.07

8. Secondary Outcome: Change From Baseline in the CGI-I Score
Description: The Clinical Global Impression - Improvement (CGI-I) Score is a clinician's impression of how much the participant's illness has improved or worsened relative to the baseline on a 7-point scale. Scores ranged from 1-7 on a scale of 1 (very much improved) to 7 (very much worse). Higher values represent a worse outcome.
Time Frame: Week 5, 8, 11, 14, 18, 22, 26, and 27
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Tavapadon 5 mg | Tavapadon 15 mg
Number analyzed (Participants) | 174 | 174 | 172
score on a scale
  Week 5: number analyzed (Participants) | 171 | 154 | 160
  Week 5 | 3.8 (0.06) | 3.4 (0.06) | 3.4 (0.06)
  Week 8: number analyzed (Participants) | 167 | 148 | 150
  Week 8 | 3.8 (0.06) | 3.2 (0.07) | 3.3 (0.07)
  Week 11: number analyzed (Participants) | 160 | 141 | 134
  Week 11 | 3.8 (0.07) | 3.0 (0.08) | 3.1 (0.08)
  Week 14: number analyzed (Participants) | 158 | 142 | 134
  Week 14 | 3.8 (0.07) | 3.0 (0.08) | 3.0 (0.08)
  Week 18: number analyzed (Participants) | 153 | 138 | 128
  Week 18 | 3.9 (0.08) | 2.8 (0.08) | 2.9 (0.08)
  Week 22: number analyzed (Participants) | 150 | 136 | 126
  Week 22 | 3.9 (0.08) | 2.9 (0.09) | 3.0 (0.09)
  Week 26: number analyzed (Participants) | 148 | 132 | 117
  Week 26 | 3.9 (0.09) | 2.8 (0.09) | 3.0 (0.09)
  Week 27: number analyzed (Participants) | 147 | 134 | 119
  Week 27 | 4.0 (0.09) | 2.8 (0.09) | 2.9 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Tavapadon 5 mg; Week 26; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -1.1, 95% CI 2-sided [-1.4 to -0.9], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Placebo vs Tavapadon 15 mg; Week 26; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -1.0, 95% CI 2-sided [-1.2 to -0.7], Standard Error of Mean 0.12

9. Secondary Outcome: Change From Baseline in the PGIC Score
Description: as for outcome 3
Time Frame: Week 5, 8, 11, 14, 18, 22, 26, and 27
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Tavapadon 5 mg | Tavapadon 15 mg
Number analyzed (Participants) | 174 | 174 | 172
score on a scale
  Week 5: number analyzed (Participants) | 171 | 155 | 160
  Week 5 | 3.7 (0.07) | 3.5 (0.07) | 3.4 (0.07)
  Week 8: number analyzed (Participants) | 168 | 148 | 151
  Week 8 | 3.8 (0.08) | 3.2 (0.08) | 3.2 (0.08)
  Week 11: number analyzed (Participants) | 161 | 141 | 135
  Week 11 | 3.8 (0.08) | 3.0 (0.08) | 3.1 (0.08)
  Week 14: number analyzed (Participants) | 159 | 142 | 134
  Week 14 | 3.8 (0.08) | 2.8 (0.09) | 3.0 (0.09)
  Week 18: number analyzed (Participants) | 154 | 137 | 129
  Week 18 | 3.9 (0.09) | 2.8 (0.10) | 2.9 (0.10)
  Week 22: number analyzed (Participants) | 151 | 137 | 126
  Week 22 | 3.8 (0.09) | 2.9 (0.10) | 2.9 (0.10)
  Week 26: number analyzed (Participants) | 147 | 132 | 117
  Week 26 | 4.0 (0.10) | 2.8 (0.10) | 2.8 (0.11)
  Week 27: number analyzed (Participants) | 147 | 134 | 119
  Week 27 | 4.0 (0.10) | 2.8 (0.11) | 2.9 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Tavapadon 5 mg; Week 26; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -1.2, 95% CI 2-sided [-1.4 to -0.9], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo vs Tavapadon 15 mg; Week 26; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -1.2, 95% CI 2-sided [-1.5 to -0.9], Standard Error of Mean 0.14

10. Secondary Outcome: Change From Baseline in the Epworth Sleepiness Scale (ESS)
Description: The ESS is an 8-question, participant questionnaire that is intended to measure daytime sleepiness. It assesses the likelihood of dozing off or falling asleep in the following common situations: sitting and reading, sitting inactive in a public place as a passenger in a car for an hour or more without stopping for a break, lying down to rest when circumstances permit, sitting and talking to someone, sitting quietly after a meal without alcohol, and in a car while stopped for a few minutes in traffic or at a light.
  Each situation is rated on a 4-point (0-3) scale with scores ranging from 0 (would never nod off) to 3 (high chance of nodding off). Higher values represent a worse outcome.
Time Frame: Week 26
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Tavapadon 5 mg | Tavapadon 15 mg
Number analyzed (Participants) | 148 | 134 | 118
score on a scale | -0.2 (0.23) | -0.3 (0.24) | -0.5 (0.24)
Statistical Analysis 1: Comparison: Placebo vs Tavapadon 5 mg; Week 26; Test type: Superiority; p = 0.6047, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.2, 95% CI 2-sided [-0.8 to 0.5], Standard Error of Mean 0.32
Statistical Analysis 2: Comparison: Placebo vs Tavapadon 15 mg; Week 26; Test type: Superiority; p = 0.2570, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.4, 95% CI 2-sided [-1.0 to 0.3], Standard Error of Mean 0.33

11. Secondary Outcome: Change From Baseline in the Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS)
Description: QUIP-RS is a questionnaire for impulse-compulsive disorders in Parkinson's disease rating scale to assess impulse control disorders (ICD). The QUIP-RS has 4 primary questions that pertain to commonly reported thoughts, urges/desires, and behaviors associated with ICDs, each of which is applied to 4 ICDs (compulsive gambling, buying, eating, sexual behavior) and 3 related disorders (medication use, punding, and hobbyism). The QUIP-RS uses a 5-point Likert scale (score 0-4 [0 means "never" and 4 means "very often"] for each question) to gauge the frequency of behaviors. Scores for each ICD and related disorder range from 0 to 16, with a higher score indicating greater severity (frequency) of symptoms. The total QUIP-RS score for all ICDs and related disorders combined ranges from 0 to 112. A higher score indicating greater severity of symptoms.
Time Frame: Week 26
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Tavapadon 5 mg | Tavapadon 15 mg
Number analyzed (Participants) | 147 | 134 | 118
score on a scale | -2.1 (0.46) | -2.2 (0.47) | -2.4 (0.48)
Statistical Analysis 1: Comparison: Placebo vs Tavapadon 5 mg; Week 26; Test type: Superiority; p = 0.8516, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.1, 95% CI 2-sided [-1.4 to 1.1], Standard Error of Mean 0.63
Statistical Analysis 2: Comparison: Placebo vs Tavapadon 15 mg; Week 26; Test type: Superiority; p = 0.6421, Mixed-effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.3, 95% CI 2-sided [-1.6 to 1.0], Standard Error of Mean 0.64

12. Secondary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a systematically administered instrument developed to track suicidal adverse events across a treatment study. The instrument is designed to assess suicidal behavior and ideation, track and assess all suicidal events, as well as the lethality of attempts. Suicidal ideation (SI) categories include the following: wish to be dead; nonspecific active suicidal thoughts; active suicidal ideation without intent to act; active suicidal ideation with some intent to act but no plan; active suicidal ideation with plan and intent. Suicidal behavior categories include the following: actual attempt; interrupted attempt; aborted attempt; preparatory acts or behavior; suicidal behavior; completed suicide.
Time Frame: Week 27
Population: Population includes subjects who received at least one dose of study drug and had available data for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tavapadon 5 mg | Tavapadon 15 mg
Number analyzed (Participants) | 175 | 177 | 177
Participants
  Participants With Any Suicidal Ideations | 3 | 3 | 3
  Participants With Any Suicidal Behaviors | 0 | 0 | 0
  Participants With Any Suicidal Behaviors or Ideations | 3 | 3 | 3
  Participants With Non-Suicidal Self-Injurious Behavior | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: From first dose of study drug until 190 days following last dose of study drug.
Population: All-treated data set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tavapadon 5 mg | Tavapadon 15 mg
Number analyzed (Participants) | 175 | 177 | 177
Participants | 100 | 142 | 139

ADVERSE EVENTS:
Time Frame: All-cause mortality was reported from enrollment until 4 weeks after the last dose of study drug. Treatment-emergent adverse events and serious adverse events were collected from the first dose of study drug until 4 weeks after the dose of study drug for all Arms. Mean duration on study drug was 27 weeks. Median time on study was 190, 190, 189 days for Placebo, Tavapadon 5 mg, and Tavapadon 15 mg, respectively.
Groups:
- Tavapadon 5mg QD: Participants will receive tavapadon tablet titrated up to 5 milligram (mg) once daily (QD) orally for 27 weeks.
- Tavapadon 15mg QD: Participants will receive tavapadon tablet titrated up to 15 milligram (mg) QD orally for 27 weeks.
Arm/Group | Placebo | Tavapadon 5mg QD | Tavapadon 15mg QD
All-Cause Mortality (participants affected / at risk) | 2/175 | 1/177 | 0/177
Serious Adverse Events (participants affected / at risk) | 11/175 | 4/177 | 10/177
Other Adverse Events (participants affected / at risk) | 72/175 | 125/177 | 125/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=175) | Tavapadon 5mg QD (N=177) | Tavapadon 15mg QD (N=177)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DEATH (General disorders) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
TRACHEOBRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
HALLUCINATION, TACTILE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=175) | Tavapadon 5mg QD (N=177) | Tavapadon 15mg QD (N=177)
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 6 (6) | 3 (3)
VERTIGO (Ear and labyrinth disorders) | 2 (2) | 5 (6) | 3 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (4)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (8)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 4 (4) | 5 (5)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (3)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 11 (12) | 9 (9)
DYSPEPSIA (Gastrointestinal disorders) | 2 (3) | 5 (6) | 10 (10)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 7 (7) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 3 (5) | 42 (44) | 48 (56)
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (4)
VOMITING (Gastrointestinal disorders) | 1 (2) | 12 (13) | 9 (11)
ASTHENIA (General disorders) | 0 (0) | 5 (5) | 2 (2)
FATIGUE (General disorders) | 6 (6) | 10 (11) | 16 (17)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 4 (5) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4) | 9 (9) | 6 (6)
NASOPHARYNGITIS (Infections and infestations) | 4 (5) | 2 (2) | 6 (6)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 0 (0) | 4 (4)
URINARY TRACT INFECTION (Infections and infestations) | 9 (10) | 6 (7) | 3 (4)
FALL (Injury, poisoning and procedural complications) | 6 (6) | 4 (4) | 7 (8)
SARS-COV-2 TEST POSITIVE (Investigations) | 2 (2) | 4 (4) | 0 (0)
WEIGHT DECREASED (Investigations) | 2 (2) | 3 (4) | 4 (4)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 5 (5)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (5) | 4 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (8) | 4 (4)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 3 (3)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4) | 4 (4)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (7) | 5 (5)
AGEUSIA (Nervous system disorders) | 0 (0) | 1 (1) | 5 (6)
DIZZINESS (Nervous system disorders) | 8 (9) | 24 (32) | 21 (23)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 14 (14) | 14 (17)
HEADACHE (Nervous system disorders) | 9 (16) | 22 (25) | 37 (39)
HYPOAESTHESIA (Nervous system disorders) | 2 (2) | 3 (4) | 6 (9)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 3 (5) | 8 (11)
PAROSMIA (Nervous system disorders) | 0 (0) | 4 (4) | 4 (4)
SOMNOLENCE (Nervous system disorders) | 6 (6) | 6 (6) | 5 (5)
TREMOR (Nervous system disorders) | 2 (3) | 4 (4) | 3 (3)
ABNORMAL DREAMS (Psychiatric disorders) | 1 (1) | 10 (10) | 6 (6)
ANXIETY (Psychiatric disorders) | 5 (5) | 10 (11) | 9 (10)
DEPRESSION (Psychiatric disorders) | 4 (4) | 2 (2) | 4 (4)
HALLUCINATION, VISUAL (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (5)
INSOMNIA (Psychiatric disorders) | 4 (4) | 5 (5) | 7 (8)
SLEEP DISORDER (Psychiatric disorders) | 1 (1) | 4 (4) | 3 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 6 (6)
HYPERTENSION (Vascular disorders) | 8 (8) | 1 (1) | 2 (2)
HYPOTENSION (Vascular disorders) | 4 (4) | 7 (9) | 8 (9)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 11 (11) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT04201093/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/93/NCT04201093/SAP_001.pdf